CLINICAL TRIAL: NCT03874637
Title: Evaluation of a Wearable Electrical Incontinence Device in Subjects: A Non-significant Risk Clinical Evaluation of FemPulse Therapy in Women With OAB
Brief Title: FemPulse Therapy First-in-Human Experience
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: FemPulse Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Other
Other Study IDs: CIP-001
Record Dates: First submitted 2019-03-04; First posted 2019-03-14 (Actual); Last update posted 2019-03-14 (Actual); Status verified 2019-02

CONDITIONS: Urinary Bladder, Overactive
Keywords: Overactive Bladder; Women; Neuromodulation; Bioelectronic Medicine; Non-significant Risk
MeSH Terms: conditions — Urinary Bladder, Overactive

STUDY DESIGN:
Intervention Model Description: Subjects will be treated at 2 different device settings (one of which is Off) in random sequence during two 6-hour periods at least one week apart.
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (2):
- Treatment (Experimental): Active therapy
  Interventions: Device: Treament
- Sham Control (Sham Comparator): Sham Control
  Interventions: Device: Sham Control

INTERVENTIONS:
Device: Treament — Placement of the FemPulse System with therapy delivery
  Arms: Treatment
Device: Sham Control — Placement of the FemPulse System without therapy delivery
  Arms: Sham Control

SUMMARY:
The purpose of this clinical trial is to investigate a new medical device treatment for Overactive Bladder (OAB) in women.

DETAILED DESCRIPTION:
The FemPulse System is a vaginal ring intended to provide mild electrical stimulation to nerves in the lower abdomen that regulate bladder function. It is believed that stimulation of these nerves may help relieve the symptoms of OAB.

ELIGIBILITY:
Inclusion Criteria:

* Females ≥21 yrs with Overactive Bladder

Exclusion Criteria:

* Is or was recently pregnant
* Has a metal pelvic implant or any electrically active implanted medical device
* Has a urinary tract or vaginal infection
* Had a previous hysterectomy, pelvic radiation or pelvic cancer
* Has significant pelvic organ prolapse
* Had bladder treatment with onabotulinumtoxinA in the previous 12 months or Tibial Nerve stimulation within the previous 30 days
* Has a significant heart condition or a history of vasovagal reaction or low blood pressure

Min Age: 21 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2017-02-14 (Actual); Primary Completion 2017-05-17 (Actual); Study Completion 2017-05-17 (Actual)

PRIMARY OUTCOMES:
Adverse Events | 3 days in total
  All device- and procedure-related adverse events will be collected and tabulated
Placeability and comfort of the device | 3 days in total
  Subjects will be observed for their ability to place, orient and wear the device without discomfort. The outcome is Pass or Fail as determined by the investigator.

SECONDARY OUTCOMES:
Frequency of urinary voids | 3 days in total
  The number of voids per day will be tabulated
Intervals between urinary voids | 3 days in total
  The time between voids (hours:minutes) will be tabulated
Urge urinary incontinence (UUI) | 3 days in total
  Presence or absence of UUI with each void

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Minnesota Urology, Woodbury, Minnesota
  - University of Washington Medical Center, Seattle, Washington

IPD SHARING:
Plan to Share IPD: No